CLINICAL TRIAL: NCT00006786
Title: Phase II Trial of Fluorouracil (5-FU), Leucovorin (LV), Irinotecan (CPT-11) and Bevacizumab (Anti-VEGF) in Previously Untreated Patients With Advanced Colorectal Cancer
Brief Title: Combination Chemotherapy Plus Bevacizumab in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068328; ECOG-E2200
Record Dates: First submitted 2000-12-06; First posted 2004-02-12 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2006-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Irinotecan; Leucovorin

INTERVENTIONS:
Biological: bevacizumab
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Bevacizumab may stop the growth of colorectal cancer by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus bevacizumab in treating patients who have advanced colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the progression-free survival at 7 months of patients with previously untreated advanced colorectal cancer treated with fluorouracil, leucovorin calcium, irinotecan, and bevacizumab. II. Determine the response rate and overall survival of this patient population treated with this regimen. III. Determine the toxicity of this treatment regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive irinotecan IV over 90 minutes, leucovorin calcium IV, and fluorouracil IV once weekly for 4 weeks. Patients also receive bevacizumab IV over 30-90 minutes once every 2 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced or metastatic adenocarcinoma of the colon and rectum Surgically unresectable disease Measurable disease Disease outside the prior radiotherapy port and/or progressive disease within the previously irradiated volume

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 No hemorrhagic events within the past 6 months Hepatic: Bilirubin normal SGOT normal INR no greater than 1.5 Renal: Creatinine no greater than 1.5 times upper limit of normal Cardiovascular: No thromboembolic events within the past 6 months Pulmonary: No evidence of pneumonia Other: No known hypersensitivity to recombinant humanized murine monoclonal antibodies No evidence of significant active infection (e.g., peritonitis or wound abscess) Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent sargramostim (GM-CSF) Chemotherapy: At least 12 months since prior fluorouracil-based adjuvant chemotherapy No prior adjuvant irinotecan Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 2 weeks since prior radiotherapy and recovered Surgery: See Disease Characteristics Other: No prior therapy for advanced disease No concurrent therapeutic anticoagulation except for low-dose coumadin for maintenance of indwelling catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J. Giantonio, MD, Study Chair — Presbyterian medical center
Locations (77):
- United States (74):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - MBCCOP-Howard University Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainsville, Gainesville, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Veterans Affairs Medical Center - Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Puerto Rico (2):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Background] Giantonio BJ, Chen HX, Catalano PJ, et al.: Bowel perforation and fistula formation in colorectal cancer patients treated on Eastern Cooperative Oncology Group (ECOG) studies E2200 and E3200. [Abstract] J Clin Oncol 22 (Suppl 14): A-3017, 199s, 2004.
- [Background] Gray R, Giantonio BJ, O'Dwyer PJ, et al.: The safety of adding angiogenesis inhibition into treatment for colorectal, breast, and lung cancer: the Eastern Cooperative Oncology Group's (ECOG) experience with bevacizumab (anti-VEGF). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-825, 2003.
- [Result] Giantonio BJ, Levy DE, O'dwyer PJ, Meropol NJ, Catalano PJ, Benson AB 3rd; Eastern Cooperative Oncology Group. A phase II study of high-dose bevacizumab in combination with irinotecan, 5-fluorouracil, leucovorin, as initial therapy for advanced colorectal cancer: results from the Eastern Cooperative Oncology Group study E2200. Ann Oncol. 2006 Sep;17(9):1399-403. doi: 10.1093/annonc/mdl161. Epub 2006 Jul 27. PMID 16873427
- [Result] Giantonio BJ, Levy D, O'Dwyer PJ, et al.: Bevacizumab (anti-VEGF) plus IFL (irinotecan, fluorouracil, leucovorin) as front-line therapy for advanced colorectal cancer (advCRC): results from the Eastern Cooperative Oncology Group (ECOG) Study E2200. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1024, 2003.
- [Result] Giantonio BJ, Levy D, Catalano PJ, et al.: Incorporating angiogenesis inhibition with bevacizumab (anti-VEGF) into frontline chemotherapy with irinotecan (CPT-11), fluorouracil and leucovorin (FU/LV) for advanced colorectal cancer (advCRC): a toxicity analysis of ECOG study E2200. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-503, 2002.